CLINICAL TRIAL: NCT03716284
Title: Electromagnetic Navigation Bronchoscopy for the Diagnosis of Peripheral Pulmonary Nodules: a Real World Study
Brief Title: ENB for the Diagnosis of PPNs:a Real World Study
Status: Completed | Type: Observational
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Air Force Military Medical University, China (Other); Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director, Department of Endoscopy, Shanghai Chest Hospital
Other Study IDs: 2017YFC0112701-2
Record Dates: First submitted 2018-10-20; First posted 2018-10-23 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Peripheral Pulmonary Nodules
Keywords: electromagnetic navigation bronchoscopy(ENB); peripheral pulmonary nodules; diagnostic yield

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Electromagnetic navigation bronchoscopy (ENB) — ENB is carried out by a ENB system（LungCare, China) with/without other guided bronchoscopy techniques and/or ROSE, which can offer real-time navigation for bronchoscopy reaching peripheral pulmonary nodules.

SUMMARY:
The study is designed as a multi-center prospective trial of ENB for the diagnosis of peripheral pulmonary nodules in the real world. The purpose of the study is to identify the optimal method of using ENB.

DETAILED DESCRIPTION:
The study will be conducted at no less than 5 clinical centers. Patients with peripheral pulmonary nodules suspicious for malignancy will be enrolled in the study. ENB will be performed with/without other guided bronchoscopy techniques and/or ROSE. Different biopsy methods will be recorded as well. The primary endpoint is the diagnostic yield of ENB. The secondary endpoints include factors affecting diagnostic yield, operation time, complications, safety and so on.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are older than 18 year-old.
2. Chest CT shows peripheral pulmonary nodule (8mm<longest diameter≤30mm) suspicious for malignant that needs to be confirmed by pathology. The nodule is surrounded by lung parenchyma and invisible with standard bronchoscopy.
3. Patients who agree to undergo bronchoscopy without any contraindications.
4. Patients who have good compliance and sign informed consent.

Exclusion Criteria:

1. Presence of concomitant endobronchial lesion during the brochoscopy procerdure.
2. Severe cardiopulmonary dysfunction and other indications that can't receive bronchoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet inclusion/exclusion criteria will be enrolled in the study consecutively in each clinical center.
Sampling Method: Probability Sample
Enrollment: 479 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield | One year
  Diagnostic yield is defined as proportion of true positive and true negative. The primary endpoint is diagnostic yield of ENB with/without other guided bronchoscopy techniques or ROSE.

SECONDARY OUTCOMES:
The difference of diagnostic yield among groups of different methods of using ENB | One year
  ENB will be performed with/without other guided bronchoscopy techniques and/or ROSE. Different biopsy methods will be recorded as well.The difference of diagnostic yield among groups of different methods of using ENB will be analyzed.
Factors affecting diagnostic yield | One year
  Factors affecting diagnostic yield including lesion size,bronchus sign, location and so on will be analyzed.
The difference of diagnostic yield among groups using different locatable guides | One year
  There are three kinds of locatable guides with different outer diameters. The difference of diagnostic yield among groups using different locatable guides will be analyzed.
Operation time | One year
  Operation time includes total operation time,total GS time and total EBUS time.
Incidence of complications | One year
  Complications mean a composite of operation-related serious adverse events (pneumothorax, bleeding, etc.) during and after the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, MD,PhD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Khandhar SJ, Bowling MR, Flandes J, Gildea TR, Hood KL, Krimsky WS, Minnich DJ, Murgu SD, Pritchett M, Toloza EM, Wahidi MM, Wolvers JJ, Folch EE; NAVIGATE Study Investigators. Electromagnetic navigation bronchoscopy to access lung lesions in 1,000 subjects: first results of the prospective, multicenter NAVIGATE study. BMC Pulm Med. 2017 Apr 11;17(1):59. doi: 10.1186/s12890-017-0403-9. PMID 28399830
- [Background] Ost DE, Ernst A, Lei X, Kovitz KL, Benzaquen S, Diaz-Mendoza J, Greenhill S, Toth J, Feller-Kopman D, Puchalski J, Baram D, Karunakara R, Jimenez CA, Filner JJ, Morice RC, Eapen GA, Michaud GC, Estrada-Y-Martin RM, Rafeq S, Grosu HB, Ray C, Gilbert CR, Yarmus LB, Simoff M; AQuIRE Bronchoscopy Registry. Diagnostic Yield and Complications of Bronchoscopy for Peripheral Lung Lesions. Results of the AQuIRE Registry. Am J Respir Crit Care Med. 2016 Jan 1;193(1):68-77. doi: 10.1164/rccm.201507-1332OC. PMID 26367186
- [Background] Folch EE, Bowling MR, Gildea TR, Hood KL, Murgu SD, Toloza EM, Wahidi MM, Williams T, Khandhar SJ. Design of a prospective, multicenter, global, cohort study of electromagnetic navigation bronchoscopy. BMC Pulm Med. 2016 Apr 26;16(1):60. doi: 10.1186/s12890-016-0228-y. PMID 27113209
- [Background] Gex G, Pralong JA, Combescure C, Seijo L, Rochat T, Soccal PM. Diagnostic yield and safety of electromagnetic navigation bronchoscopy for lung nodules: a systematic review and meta-analysis. Respiration. 2014;87(2):165-76. doi: 10.1159/000355710. Epub 2014 Jan 3. PMID 24401166
- [Derived] Li Y, Chen W, Xie F, Huang R, Liu X, Xiao Y, Cao L, Hu Y, Ke M, Wu S, Sun J. Novel electromagnetic navigation bronchoscopy system for the diagnosis of peripheral pulmonary nodules: a prospective, multicentre study. Thorax. 2023 Dec;78(12):1197-1205. doi: 10.1136/thorax-2022-219664. Epub 2023 Sep 21. PMID 37734951
- [Derived] Jiang S, Liu X, Chen J, Ma H, Xie F, Sun J. A pilot study of the ultrathin cryoprobe in the diagnosis of peripheral pulmonary ground-glass opacity lesions. Transl Lung Cancer Res. 2020 Oct;9(5):1963-1973. doi: 10.21037/tlcr-20-957. PMID 33209616